CLINICAL TRIAL: NCT02446977
Title: Randomized Clinical Trial to Investigate Whether Administration of CBG000592 (Riboflavin/Vitamin B2) in Patients With Acute Ischemic Stroke Causes a Reduction of Glutamate-mediated Excitotoxicity
Brief Title: Administration of CBG000592 (Riboflavin/Vitamin B2) in Patients With Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Castillo, José, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JCS-CBG-2014-01; NCT02540980 (obsolete NCT alias)
Record Dates: First submitted 2015-04-21; First posted 2015-05-18 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Ischemic Stroke
Keywords: ischemic; stroke; vitamin B2
MeSH Terms: conditions — Ischemic Stroke; Ischemia; Stroke | interventions — Solutions; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin B2 Streuli® (Experimental): 20mg IV
  Interventions: Drug: Vitamin B2 Streuli®
- Solution for injection (Placebo Comparator): 4ml IV
  Interventions: Other: Solution for injection

INTERVENTIONS:
Drug: Vitamin B2 Streuli® — 4ml IV
  Other Names: CBG000592
  Arms: Vitamin B2 Streuli®
Other: Solution for injection — 4ml IV
  Other Names: Placebo Comparator
  Arms: Solution for injection

SUMMARY:
Administration of CBG000592 (riboflavin/vitamin B2) in patients with acute ischemic stroke to know if it causes a reduction of glutamate-mediated excitotoxicity.

DETAILED DESCRIPTION:
The investigators hypothesis focuses on the effect of riboflavin given for the first three hours of ischemic stroke, as a reducing agent of cerebral glutamate concentration. This administration would produce a reduction of excitotoxic damage and consequently generate clinical improvement, while a lower income and a better functional outcome of patients at three months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years, both men and women.
2. Patient or legal representative able to understand and sign the informed consent.
3. Patients with suspected stroke within 3 hours of onset.

Exclusion Criteria:

1. Women of childbearing age, with potential for pregnancy or breastfeeding.
2. Patients with a score ≥ 2 point 1a in the NIHSS scale.
3. Scale pre-stroke modified Rankin ≥ 2.
4. Inability to prior testing image needed for the study.
5. Previous disorders that may interfere with the interpretation of neurological scales.
6. Treatment with probenecid, tricyclic antidepressants, phenothiazines, streptomycin, erythromycin, tyrothricin, tetracyclines and carbomycin, at the time of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reduction of serum glutamate concentration | 7 hours
  Difference between serum glutamate concentration from basal (prior to medication infusion) and levels at 3 ± 1 and 6 ± 1 hours, from administered medication, including branch CBG000592 (riboflavin/vitamin B2) and placebo.

SECONDARY OUTCOMES:
Days of hospitalisation | 3 months
  To study the average length of stay in patients with acute ischemic stroke: difference in days, between patient arrival and the patient's discharge, between the two treatment arms.
Percentage of clinical improvement (basal-high) | 3 months
  To study the rate of clinical improvement in patients with acute ischemic stroke: clinical improvement according to the formula: (NIHSSbasal-NIHSSalta) / NIHSSbasal x 100 and compared between the two treatment arms.
Functional outcome using Rankin Scale at 90 days | 3 months
  Study the functional outcome in patients with acute ischemic stroke: modified Rankin scale at 90 days, between two treatment arms.
Serum glutamate concentrations | 7 hours
  Variations of serum glutamate curves in patients with acute ischemic stroke between two branches: all concentrations of serum glutamate.
Prognosis of patients using Rankin Scale at 90 days | 3 months
  To explore the prognosis of patients without stroke, evaluating modified Rankin scale at 90 days.
Number of participants with Adverse Event | 3 months
  Safety management: measuring adverse events throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: José Castillo, MD, Study Director — Complejo Hospitalario Universitario de Santiago
Locations (1):
- Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña, Spain